CLINICAL TRIAL: NCT01554787
Title: Randomized, Double Blind, Placebo Control Trial to Evaluate the Efficacy of Astragalus Membranaceus in the Patients After Stroke With Fatigue
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMR100-IRB-251
Record Dates: First submitted 2012-03-07; First posted 2012-03-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Fatigue; Stroke
Keywords: After stroke with fatigue
MeSH Terms: conditions — Fatigue; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Chinese Herb Astragalus membranaceus (Experimental)
  Interventions: Drug: Chinese Herb Astragalus membranaceus
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Chinese Herb Astragalus membranaceus — Astragalus membranaceus(AM)at a rate of 2.8g three times per day
  Arms: Chinese Herb Astragalus membranaceus
Other: Placebo — at a rate of 2.8g three times per day
  Arms: Placebo

SUMMARY:
The high levels of fatigue in stroke patients without neurological impairment suggest it has a central origin rather than being the result of increased physical effort required after stroke（Winward et al., 2009）. Fatigue is different from post-stroke depression and the more serious stroke patients are more prone to fatigue（Windward et al., 2009）.

Fatigue is one of the symptoms of qi deficiency,and Astragalus membranaceus is the most effective of all traditional Chinese medicine and can tonifying middle and tonify the original qi. Therefore, the aim of this study was to investigate the efficacy of Astragalus membranaceus on post-stroke fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Male or female.
2. Age: between 40 and 80 years old.
3. Three months after stroke.
4. Hemorrhagic stroke or ischemic stroke.
5. Fatigue score from screen process ≧4.
6. Subject with comprehension or communication.
7. Volunteer signs the agreement to participate the study after whole study purpose and procedures description in detail.

Exclusion Criteria:

1. People from mental illness can not to participate the evaluation.
2. Major diseases such as cancer、Chronic pulmonary obstructive disease(COPD)、 Heart failure、Myocardial Infraction、Chronic renal failure or Liver cirrhosis.
3. Pregnant woman.
4. Breast-feeding woman.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ-C30 | 2 year(all patients)
BFI-T score | 2 years(all patients)

SECONDARY OUTCOMES:
SF-36 score | 2 years(all patients)

CONTACTS AND LOCATIONS:
Overall Officials: Chung Hsiang Liu, MD., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan